CLINICAL TRIAL: NCT05412537
Title: The Impact of Motivation in Return to Work After Work Disability
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: S62188
Record Dates: First submitted 2020-11-09; First posted 2022-06-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Motivation; Quality of Life; Communication; Health Behavior
MeSH Terms: conditions — Communication; Health Behavior

STUDY DESIGN:
Intervention Model Description: The RCT will compare two groups: (a) a consult as usual (a regular consult with the medical advisor) and (b) an intervention based on motivational interviewing performed by a medical advisor.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAU (Active Comparator): A sickness funds provides a physician or paramedic's consultation with people on work disability 3 to 6 months after the onset of the sickness period. The goal of this conversation is (1) to gather information on the reason of work disability, (2) gather information of the treatment plan and (3) to encourage people to RTW.
  CAU stands for consult as usual
  Interventions: Other: CAU
- Motivational Interviewing (Experimental): Motivational Interviewing involves a conversation about behavioral change in terms of recovery or RTW. The role of the MI practitioner is to evoke change talk. By change talk, the patient expresses a desire, a reason, an ability or a need for change. It is of importance that patients themselves generate the motivation for change, and it is the practitioner's task to assist them in making informed and contemplated choices to act. The core idea is that people have to become motivated themselves to change such that the new behavior is something that they want instead of something that someone else wants. There are 4 processes: engaging, focusing, evoking and planning. Training in MI for health care professionals typically is provided in 1- to 3-day workshops. This is consistent with the 2-day training in the current research. MI was planned 3 to 6 months after the onset of work disability.
  Interventions: Other: MI

INTERVENTIONS:
Other: MI — How to motivate people
  Arms: Motivational Interviewing
Other: CAU — consult as usual
  Arms: CAU

SUMMARY:
The current research on the impact of motivation in return to work after work disability has 2 major parts: (1) a questionnaire study for which SMEC gave approval, this part is completed, (2) a RCT.

The RCT will compare two groups: (a) a consult as usual (a regular consult with the medical advisor) and (b) an intervention based on motivational interviewing performed by a medical advisor.

DETAILED DESCRIPTION:
Work disability is a major rising problem and brings a high societal cost in European countries. The Belgian institute for public health insurance reported that costs for work disability for the first time have overgrown the costs of unemployment.

Work disability can be assessed in many ways. For a long time, a biomedical framework was used with focus on physiopathology. According to this framework, complaints and disability result from observable damage in the body (e.g., virus, fracture, lesion, etc.). Once damage is resolved, a patient is expected to resume activities and, for instance, return to work. In some cases, it is obvious that the patient is not able to work (e.g. a roofer with a broken leg) or is prohibited to resume work (e.g. a bus driver with a driving ban after an epileptic seizure). But how can the investigators explain the phenomenon that in two patients with similar pathology and complaints, the first one returns to work and the other does not? This requires a shift from a biomedical to a biopsychological perspective. The latter assumes a complex interplay between biological, psychological and even social factors on disease. A plentiful of psychological constructs have been studied in order to explain the observed heterogeneity on human suffering in the context of chronic diseases. One of these is the construct of motivation.

The research on motivation in the domain of psychology is on the rise. Binary thinking on motivation (being motivated or not) has been left behind since the introduction of intrinsic and extrinsic motivation in the 1970's by Edward Deci and Richard Ryan in their Self-Determination Theory (SDT). The SDT has been developed in the past 40 years based on scientific research and has been applied in various fields. Relatively recently this theory has been introduced to the work context and its usefulness has been proven. Research of the theory applied to the context of work disability is however still scarce.

Whereas other theories mainly look at how strongly people are motivated (a quantitative approach), the SDT emphasizes to look at the quality of this motivation. SDT suggests that higher levels of motivation do not necessarily yield more desirable outcomes if the motivation is of poor quality. The differences in the quality of motivation are associated with the regulation of the behavior being autonomous or controlled. Several studies confirm that both employees and unemployed feel better and how more desirable behaviors (e.g., search behavior, performance, helping) when having a more autonomous regulation and a less controlled regulation. For disabled, research showed that motivation can be improved through interventions helping to formulate realistic goals and empowering them to be responsible for their own participation despite their limitations. Autonomous regulation can be elicited by the individual self or by the environment by meeting the individual's basic psychological needs. SDT considers three needs as basic: the need for autonomy, need for belongingness and need for competence.

SDT is a theory that helps to understand how and why people get motivated. A framework that arose from practice and shares large similarities with SDT is Motivational Interviewing (MI). It consists of principles and techniques that are applied in order to increase client autonomy. Clients themselves generate the motivation for change, and it is a counselor's task to help clients detect ambivalence regarding behavior change, and assist them in making informed and contemplated choices to act. MI has been proven an effective approach to promote behavioral change and may therefore be especially beneficial in a RWT context as returning to work can be conceptualized as a complex human behavior change, involving physical recovery, motivation, behavior, etc. It was found that MI, in addition to routine functional restoration, is more effective than a routine functional restoration program alone in improving RTW among workers with disabling musculoskeletal disorders. Research furthermore suggested that MI may be an effective method to facilitate RTW. SDT may prove to be a useful theoretical model to understand how and why MI works within the context of RTW.

The general objective of this dissertation is to examine how motivation impacts RTW after work disability. The investigators are focusing on the question of whether motivation can be measured, and if so, whether the differences in motivation have an impact on RTW. Subsequently the question rose whether the investigators can influence motivation regarding RTW. The following research questions were investigated:

The RCT will compare two groups: (a) a consult as usual (a regular consult with the medical advisor) and (b) an intervention based on motivational interviewing performed by a medical advisor.

* the investigators suppose that a more controlled regulation, less autonomous motivation or amotivation is associated to worse or later RTW rates or RTW behavior.
* the investigators expect a lower quality of life, lower workabilty and less satisfaction in the CAU compared to MI
* the investigators are assuming that we can influence the quality of motivation within the group of work disabled people by applying Motivational Interviewing during the consultations.
* the investigators assume better progress in motivation for people with controlled motivation compared to people with amotivation or autonomous motivation
* the investigators expect worse return to work rates after 6 months for the CAU compared to MI

ELIGIBILITY:
Inclusion Criteria:

* speak and understand Dutch
* work disabled for longer than a month

Exclusion Criteria:

* work disabled for shorter dan 1 month or longer than 1 year
* not having the mental capabilities to understand the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Return to work rates | 6 months
  How many people have (partially) returned to work

SECONDARY OUTCOMES:
Quality of life SF36v2 | 3 months
  Quality of life was measured by the EQ-5D-5L. The EQ-5D is the most well-known and commonly used generic measure of health status internationally. The 5L version appears to be a valid extension of the 3-level system. The EQ-5D-5Lt is a brief self-reported questionnaire on current health and consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each of the dimensions has 3 levels of functioning: no problems, some problems, and unable to/extreme problems.Quality of life was measured at baseline and 3 months after the intervention.
Workability index | 3 months
  The single-item question on work ability (Ahlstrom, Grimby-Ekman, Hagberg, & Dellve, 2010) was used in the current research, since research shows a very strong association between the Work Ability Index (WAI; 10 items) and the single-item question. The WAI is a tool designed for occupational health services and is used today in practice as well as in research in order to assess work ability. In this study, the single-item question concerned the WAI item "current work ability compared with the lifetime best", with a possible score of 0 ("completely unable to work") to 10 ("work ability at its best"). Workability was measured at baseline, 1 week and 3 months after the intervention.
motivation for work | 3 months
  The Motivation at work scale (MAWS; Gagné, Forest, Vansteenkiste, et al., 2014) is a tool to measure controlled motivation, autonomous motivation and amotivation. Participants were asked about their motivation for their latest or current job (before their work disability). Responses were made on a seven-point scale from 1 (strongly disagree) to 7 (totally agree). Controlled motivation was measured by summing up the subscales of external and introjected motivation. Autonomous motivation was measured by summing up identified and intrinsic motivation. Amotivation was rated as a separate scale. Motivation was measured at baseline and 3 months after the intervention.
basic psychological needs | 1 week and 3 months
  The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS; Chen, Vansteenkiste, Beyers, et al., 2014) is a tool to assess basic psychological need satisfaction and basic psychological need frustration. Responses were made on a five-point scale from 1 (strongly disagree) to 5 (totally agree). Need satisfaction was measured by summing up the subscales of autonomy satisfaction, relatedness satisfaction and competence satisfaction. Need frustration was measured by summing up the subscales of autonomy frustration, relatedness frustration and competence frustration. The BPNSFS was measured at baseline, 1 week and 3 months after the intervention.
subjective experiences of the consult | 1 week and 3 months
  The patients were asked to rate their conversation based on 6 questions: (1) The conversation with the doctor/paramedic has had a positive influence on the feeling to be more in control of my recovery; (2) The conversation with the doctor/paramedic has had a positive influence on the fact that I am now taking steps in my treatment; (3) The conversation with the doctor/ paramedic has had a positive effect on my family life; (4) The conversation with the physician/paramedic has had a positive influence on my self-confidence or self-image; (5) The conversation with the physician/paramedic has had a positive influence on my perspectives on work in the long term; (6) The conversation with the doctor/paramedic has had a positive influence on my perspectives on work in the short term. Responses were made on a five-point scale from 1 (strongly disagree) to 5 (totally agree). There was room for an open answer in addition to the score they gave.
self-efficacy | 1 week and 3 months
  The Dutch general self-efficacy scale is a translated version of the general self-efficacy scale (Schwarzer & Jerusalem,1995) and measures how a person thinks and handles in general based on 10 questions. The items are scored on a four-point scale, where 1 equals "completely incorrect" and 4 corresponds to "completely correct." Self-efficacy was measured at baseline, 1 week and 3 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Du Bois, Prof. dr., Principal Investigator — KU Leuven Environment and Health
Locations (1):
- KULeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rymenans I, Vanovenberghe C, Du Bois M, Van den Broeck A, Lauwerier E. Process Evaluation of a Motivational Interviewing Intervention in a Social Security Setting: A Qualitative Study among Work-Disabled Patients. J Occup Rehabil. 2024 Mar;34(1):141-156. doi: 10.1007/s10926-023-10108-4. Epub 2023 Apr 2. PMID 37009926